CLINICAL TRIAL: NCT06450782
Title: The Effect of Post-Isometric Relaxation Technique and Myofascial Relaxation Technique on Muscle Stiffness and Pain in Individuals With Bruxism
Brief Title: The Effect of PIR and MRT on Muscle Stiffness and Pain in Individuals With Bruxism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Yunus Emre Tutuneken, Principal Investigator, Istinye University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13
Record Dates: First submitted 2024-06-05; First posted 2024-06-10 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Bruxism; Post-isometric Relaxation Technique; Myofascial Release Technique
MeSH Terms: conditions — Bruxism | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PIR Group (Experimental): Participants in the PIR Group will apply one session of post-isometric relaxation technique.
  Interventions: Other: Post-isometric Relaxation Technique; Other: Control
- MR Grup (Experimental): Participants in the MR Group will apply one session of myofascial release technique.
  Interventions: Other: Myofascial Release Technique
- Control Group (No Intervention): No intervention will be made to the participants in the Control Group.

INTERVENTIONS:
Other: Post-isometric Relaxation Technique — Sternocleidomastoid muscle Participants are asked to stretch their necks in a spuni position and then turn their heads as far to the side of the target muscle (right side) as possible until a sensation occurs that causes discomfort in the targeted SCM. In this case, the participants are asked to moderately isometrically contract the SKM muscle for 5 seconds and then relax for 3 seconds and the cervical spine is moved to the new barrier.
  Masseter muscle Participants are positioned in a sitting position. The jaw is opened as wide as possible. The index and middle fingers of one hand are placed over the lower teeth. The weight of the hand is allowed to provide flexion and traction is applied directly to the midline. In this case, the participants are asked to moderately isometrically contract the bilateral masseter muscles for 5 seconds, then relax for 3 seconds and the participant moves his chin to the new barrier.
  Arms: PIR Group
Other: Myofascial Release Technique — Sternocleidomastoid muscle The head is slightly elevated with the help of a folded towel to prevent discomfort that may develop depending on the position. The researcher sits in a chair next to the participant's head. The chair is placed at approximately 45° to the participant's neck. The participant's head is rotated 30° towards the opposite side of the treated side. The Graston instrument contacts the upper part of the SCM approximately 2 cm below the mastoid process.
  Masseter muscle It works both ways. The Graston instrument is placed on the zygomatic process of the temporal bone, approximately 1 cm in front of the ear. The soft tissue is pressed until the bone is contacted. This connection with the periosteum is maintained and a lower tension line is created towards the mandible angle. This line of tension is continued up to the mandible, where the periosteum also comes into play. It is repeated several times.
  Arms: MR Grup
Other: Control — Participants will rest for thirty minutes.
  Arms: PIR Group

SUMMARY:
Bruxism is a repetitive jaw muscle activity that occurs during sleep or while awake, characterized by teeth clenching or grinding. Bruxism affects millions of people worldwide and is considered one of the most harmful activities for the stomatognathic system due to its morphological, pathophysiological, psychosocial features and clinical consequences. Repetitive teeth clenching and grinding movements can cause spasms, stiffness, pain, and activity changes in the chewing muscles. Since bruxism is a disorder that depends on many variables, there is no single, specific treatment and multidisciplinary approaches are often required. Most treatment strategies are conservative and symptomatic, aiming to prevent the consequences of the disorder. The main purpose of physiotherapy techniques is to reduce the negative effects of bruxism on the chewing system. Physiotherapy techniques include exercises, manual therapy, electrotherapy, acupuncture, and posture awareness. It is not clear in the literature which physiotherapy techniques are effective in the management of bruxism; Therefore, more controlled studies need to be conducted. When studies in the literature are examined, no studies have been found that objectively investigate the effectiveness of relaxation techniques alone in people with muscle pain and increased muscle stiffness due to teeth clenching problems. Within the scope of this project, it is planned to investigate the effectiveness of the myofascial release technique (MRT) and post-isometric relaxation technique (PİRT) using the grastone tool.

DETAILED DESCRIPTION:
Bruxism is a repetitive jaw muscle activity that occurs during sleep or while awake, characterized by teeth clenching or grinding. Bruxism affects millions of people worldwide and is considered one of the most harmful activities for the stomatognathic system due to its morphological, pathophysiological, psychosocial features and clinical consequences. Repetitive teeth clenching and grinding movements can cause spasms, stiffness, pain, and activity changes in the chewing muscles. Since bruxism is a disorder that depends on many variables, there is no single, specific treatment and multidisciplinary approaches are often required. Most treatment strategies are conservative and symptomatic, aiming to prevent the consequences of the disorder. The main purpose of physiotherapy techniques is to reduce the negative effects of bruxism on the chewing system. Physiotherapy techniques include exercises, manual therapy, electrotherapy, acupuncture, and posture awareness. It is not clear in the literature which physiotherapy techniques are effective in the management of bruxism; Therefore, more controlled studies need to be conducted. When studies in the literature are examined, no studies have been found that objectively investigate the effectiveness of relaxation techniques alone in people with muscle pain and increased muscle stiffness due to teeth clenching problems. Within the scope of this project, it is planned to investigate the effectiveness of the myofascial release technique (MGT) and post-isometric relaxation technique (PGT) using the grastone tool. MGT provides pain relief and functional recovery by creating a low load and long-term stretching effect on the myofascial structure. Post-isometric relaxation technique (PGT), a muscle energy technique, involves voluntary contraction in a precisely controlled direction against resistance. The results of this study will reveal the effects of MGT and PGT, which have different mechanisms of action, on muscle stiffness and pain in people with bruxism. In addition, by analyzing and presenting the data obtained, the gap in the current literature will be filled and it will contribute to becoming a component of the frequently used physiotherapy program in the management of bruxism. It is expected that patients' quality of life and productivity will increase depending on the relief of their symptoms. The study is a prospective, randomized, controlled, double-blind study. People with bruxism will be informed about the study and an informed consent form will be obtained. Participants' age, gender, body weight, height and Body Mass Index (BMI) will be evaluated and recorded with a specially prepared evaluation form. Individuals with bruxism between the ages of 18-65 who volunteer to participate in the study will be included. The study included patients with neurological, psychiatric, or systemic disease, dental treatment or physical therapy, using occlusal splints, being pregnant and having active cancer, having surgery planned for the relevant areas, having no more than two molars, using removable prostheses, and those using temporomandibular joint in the last three months. People receiving treatment will be excluded. Participants will be randomly divided into three groups. Participants will be assigned to the MGT group, PGT group, and Control group. In our study, MyotonPRO will be used to evaluate the stiffness of the sternocleidomastoid and masseter muscles of bruxism patients and the visual analog scale will be used to evaluate pain. All evaluations will be made by the same researcher before and immediately after the single-session intervention. No intervention will be made to the chin and cervical area before the first measurement. There will be a 2-minute break before the second evaluation begins.

ELIGIBILITY:
Inclusion Criteria:

Being diagnosed with bruxism Being willing and volunteer to work

Exclusion Criteria:

Having a neurological, psychiatric or systemic disease Being addicted to alcohol and drugs Getting dental treatment or physical therapy Using an occlusal splint being pregnant actively having cancer Planning surgery for relevant areas Not having more than two molars Using removable dentures Receiving treatment for the temporomandibular joint in the last three months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Muscle Stiffness | 1 Day
  MyotonPRO (Muomeetria Ltd., Tallinn, Estonia) will be used to measure the stiffness of the muscles. This device works by producing a mechanical impulse on the skin over the muscle being measured. Mechanical oscillations of muscles created by mechanical impulses are measured by MyotonPRO. Muscle stiffness is measured in Newtons per meter (N/m). This method can determine the muscle's resistance to deforming forces or muscle stiffness.
  In the study, measurements will be made at room temperature at approximately 25°C, and after the participants sit on a chair for 5 minutes. During the measurement, participants will be asked to contact the SCM and masseter muscles with maximum force, and the most prominent location of the muscles will be marked. The stiffness of both muscles will be measured in both relaxed and maximum contraction conditions. All measurements will be taken 3 times and their averages will be calculated.
Pain Intensity | 1 Day
  For pain intensity according to VAS, "no pain" is usually rated as 0 points and "worst pain imaginable" as 10 points (10 cm scale). Ranges for pain intensity; <3 is mild pain, 3-6 is moderate pain, >6 is severe pain.

SECONDARY OUTCOMES:
Range Of Montion | 1 Day
  A caliper will be used for maximum mouth opening and a linear ruler will be used for slides. For maximal mouth opening, the patient will be asked to open his mouth as much as he can, the movement is repeated three times, and when the mouth is opened for the third time, the distance between the lower and upper incisors will be measured and recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Yunus Emre TÜTÜNEKEN, Istanbul, Zeytinburnu, Turkey (Türkiye)